CLINICAL TRIAL: NCT01756963
Title: Diet and Disease Activity in Patients With Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Wageningen University (Other)
Responsible Party: Sponsor
Other Study IDs: NL 42101.068.12
Record Dates: First submitted 2012-12-20; First posted 2012-12-28 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IBD-SL cohort

SUMMARY:
In addition to a genetic susceptibility, the immune system and the intestinal microbiota, diet is hypothesized to be an important factor in the onset and progression of Inflammatory Bowel Diseases (IBD). Further insight in factors affecting disease activity may contribute to targeted interventions improving disease burden and healthcare costs for these patients. However, well-designed studies exploring the role of diet in the development of exacerbations are hardly available.

The investigators hypothesize that differences in dietary patterns affects the intestinal microbiota composition and thereby contributes to the development of exacerbations in IBD.

Furthermore, a subgroup of patients suffers from malnutrition, although the exact prevalence is unknown since simple noninvasive screening tools have not been validated for IBD. The investigators hypothesize that malnutrition is frequently present in IBD patients and associated with dietary intake and disease characteristics.

ELIGIBILITY:
Inclusion Criteria:

* IBD patients, diagnosis based on clinical, endoscopic, histological and/or radiological criteria
* participating IBD-SL cohort

Exclusion Criteria:

* Unable to provide informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive IBD patients, visiting the gastroenterology outpatient clinic, participating the IBD-SL cohort
Sampling Method: Non-Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2012-11; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
The primary aim is to study the association of dietary patterns with disease activity in a consecutive cohort of IBD outpatients | 2 years

SECONDARY OUTCOMES:
To characterize intestinal microbiota in IBD patients with different dietary patterns | 2 years
To characterize the intestinal microbiota in IBD patients in remission developing an exacerbation during follow up | 2 years
To investigate the stability of the intestinal microbiota in IBD patients remaining in remission during one year follow-up | 2 years
To study the prevalence of malnutrition in a consecutive cohort of IBD outpatients | 1 year
  In a subpopulation of the present cohort (n=300) the nutritional status will be investigated
The study the association of disease characteristics and dietary intake with the prevalence of malnutrition in a consecutive cohort of IBD outpatients | 1 year
To study the sensitivity and specificity of the SNAQ / MST as malnutrition screening tool in IBD outpatients based | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: M. Pierik, MD. PhD., Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Division of Gastroenterology/Hepatology, Maastricht, Limburg, Netherlands